CLINICAL TRIAL: NCT04217421
Title: Cerebrum and Cardiac Protection With Allopurinol in Neonates With Critical Congenital Heart Disease Requiring Cardiac Surgery With Cardiopulmonary Bypass
Acronym: CRUCIAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: dr. M.J.N.L. Benders (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other); University Medical Center Nijmegen (Other); ACE Pharmaceuticals BV (Other)
Responsible Party: Sponsor-Investigator, dr. M.J.N.L. Benders, Professor, Head of Neonatology, MD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC UMCU 18-791; 2017-004596-31 (EudraCT Number)
Record Dates: First submitted 2019-11-12; First posted 2020-01-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease in Children; Neuroprotection
Keywords: Congenital Heart Disease; Neuroprotection; Allopurinol; Brain injury; Cardiopulmonary bypass; Brain function; Brain oxygenation; Cardiac function; Neurodevelopmental outcome; Cardiac surgery; Hypoxic-ischemic brain injury; Neonates
MeSH Terms: conditions — Heart Defects, Congenital; Brain Injuries; Hypoxia-Ischemia, Brain | interventions — Allopurinol; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol powder for solution for infusion (PFI) 20 mg/kg body weight per administration will be administered early postnatally (within 45 minutes and 12 hours after the first dose), preoperatively (12 hours before surgery), intraoperatively (during surgery) and postoperatively (24 hours after surgery) to the neonate in case of a prenatal CCHD diagnosis. Allopurinol PFI will be administered only pre-, intra- and postoperatively to the neonate in case of a postnatal CCHD diagnosis.
  Arms: Allopurinol
Drug: Mannitol — Mannitol powder for solution (PFI) placebo will be administered early postnatally (within 45 minutes and 12 hours after birth), preoperatively (12 hours before surgery), intraoperatively (during surgery), and postoperatively (24 hours after surgery) to the neonate in case of a prenatal CCHD diagnosis. Mannitol PFI-placebo will be administered only pre-, intra- and postoperatively to the neonate in case of a postnatal CCHD diagnosis.
  Arms: Placebo

SUMMARY:
Neurodevelopmental impairment due to delayed brain development and brain injury is a fundamental problem in children with critical congenital heart disease (CCHD). Significant longterm motor-, cognitive-, and behavioral problems are the result of early postnatally and perioperatively induced brain injury. Allopurinol, a xanthine oxidase inhibitor, prevents the formation of toxic free oxygen radicals, thereby limiting hypoxia-reperfusion damage. Both animal and neonatal studies suggest that administration of allopurinol reduces hypoxic-ischemic brain injury, is cardioprotective, and safe. This study aims to evaluate the efficacy and safety of allopurinol administered early postnatally and perioperatively in children with a CCHD requiring cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with a prenatally or postnatally confirmed diagnosis of CCHD requiring (anticipated) cardiac surgery with CPB within the first 4 weeks of life.
* Informed consent provided by both parents.

Exclusion Criteria:

* Inability to enroll the patient before the start of delivery in case of prenatal diagnosis, or 24 hours before surgery in case of postnatal diagnosis.
* Doubt whether the aortic arch anomaly before birth requires cardiac surgery with CPB in the neonatal period.
* Gestational age below 36 weeks and/or birth weight less than 2000 gram.
* Surgery not requiring cardiopulmonary bypass.
* Decision for "comfort care only".

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relevant parenchymatous brain injury on postoperative MRI | between birth and 1 month after cardiac surgery
  The presence or absence of relevant (moderate/severe) parenchymatous (ischemic or hemorrhagic) brain injury on postoperative MRI will be assessed, using the T1/T2/DWI and SWI weighted images.
Rate of children that are considered 'too unstable for postoperative MRI' | between birth and 1 month after cardiac surgery
  This decision is based on the circulatory and respiratory status of the child before the planned postoperative MRI, as included in local guidelines (not part of this protocol) of each participating center.
Incidence of mortality | between birth and 1 month after cardiac surgery
  Defined as death until one month postoperatively.

SECONDARY OUTCOMES:
Brain injury severity score on pre- and postoperative MRI | between birth and 1 month after cardiac surgery
  An MRI score, which includes diffusion-weighted imaging as well as assessment of the deep grey matter, white matter, and cerebellum [Weeke L, et al. J Pediatr 2018]. The score will be compared between groups (allopurinol vs placebo).
Volume of hypoxic-ischemic brain injury on pre- and postoperative MRI | between birth and 1 month after cardiac surgery
  To assess whether there are differences between groups (allopurinol vs placebo) in volume (mm3) of hypoxic-ischemic brain lesions using a fully automatic method for detection and quantification of ischemic lesions in diffusion-weighted MR images [Murphy K, et al. Neuroimage Clin 2017].
Global ventricular function (normal, mildly, moderately, severely, reduced) pre- and postoperatively | between birth and 1 month after cardiac surgery
Ventricular ejection fraction (%) pre- and postoperatively | between birth and 1 month after cardiac surgery
Brain function: Seizure activity on aEEG (presence or absence) postnatally and postoperatively | 24-36 hours after birth, 6 hours before surgery, 48-72 hours after surgery
Brain oxygenation: Regional cerebral oxygen saturation (%) postnatally and postoperatively | 24-36 hours after birth, 6 hours before surgery, 48-72 hours after surgery
General movements and motor optimality score | at 3 months
  Video recordings will be analyzed following the global general movement categories (normal, poor repertoire, cramped-synchronized, or chaotic) and the motor optimality score [Einspieler C, et al. Dev Med Child Neurol. 2016]. A higher score expresses a more optimal performance. Scores will be compared between groups (allopurinol vs placebo).
Neurodevelopment | at 24 months
  To assess motor, cognitive, speech and language development using the Bayley Scales of Infant and Toddler Development - Third Edition - NL (Bayley-III-NL). An average Bayley-III-NL score is 100, one standard deviation (SD) above or below the mean concerns 15 points. Scores will be compared between groups (allopurinol vs placebo).
Quality of Life (scores and subscores): TNO-AZL TAPQoL | at 24 months
  The TNO-AZL Questionnaire for Preschool Children's Health-Related Quality of Life (TAPQoL) will be assessed to give insight in the quality of life of both children with CCHD and their parents. A higher score indicates a better quality of life. Scores will be compared between groups (allopurinol vs placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Manon JNL Benders, Prof. MD PhD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht); Johannes (Hans) MPJ Breur, MD PhD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht); Nicolaas (Koos) JG Jansen, MD PhD, Study Director — University Medical Center Utrecht (UMC Utrecht); Raymond Stegeman, MD, Study Director — University Medical Center Utrecht (UMC Utrecht)
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud University Medical Center Nijmegen (Radboudumc), Nijmegen
  - Erasmus Medical Center Rotterdam (Erasmus MC), Rotterdam
  - University Medical Center Utrecht (UMC Utrecht), Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stegeman R, Nijman M, Breur JMPJ, Groenendaal F, Haas F, Derks JB, Nijman J, van Beynum IM, Taverne YJHJ, Bogers AJJC, Helbing WA, de Boode WP, Bos AF, Berger RMF, Accord RE, Roes KCB, de Wit GA, Jansen NJG, Benders MJNL; CRUCIAL trial consortium. CeRebrUm and CardIac Protection with ALlopurinol in Neonates with Critical Congenital Heart Disease Requiring Cardiac Surgery with Cardiopulmonary Bypass (CRUCIAL): study protocol of a phase III, randomized, quadruple-blinded, placebo-controlled, Dutch multicenter trial. Trials. 2022 Feb 23;23(1):174. doi: 10.1186/s13063-022-06098-y. PMID 35197082